CLINICAL TRIAL: NCT00976183
Title: A Phase I/II, Open-Label, Non-Randomized, Pilot Study of Weekly Paclitaxel, Every Four-week Carboplatin and Oral Vorinostat for Patients Newly Diagnosed With Stage III/IV Epithelial Ovarian, Fallopian Tube or Peritoneal Cancer
Brief Title: Paclitaxel, Carboplatin and Vorinostat for the Treatment of Advanced Stage Ovarian Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: toxicities
Sponsor: Gynecologic Oncology Associates (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOA-TCOV
Record Dates: First submitted 2009-09-10; First posted 2009-09-14 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2016-08

CONDITIONS: Ovarian Neoplasms
Keywords: ovarian cancer; gynecologic oncology; vorinostat; treatment
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vorinostat (Experimental): All study patients will receive the indicated dose of Vorinostat in conjunction with paclitaxel and carboplatin.
  Interventions: Drug: Vorinostat

INTERVENTIONS:
Drug: Vorinostat — Vorinostat will start at 200 mg QD on weeks 1 and 3, and escalating to 300 mg QD after safety has been evaluated following 2 cycles of treatment. If safety is acceptable, then the following patients could be treated at 400 mg QD on weeks 1 and 3.
  Other Names: suberoylanilide hydroxamic acid (SAHA)
Drug: Vorinostat — Vorinostat will be given as a lead-in dose escalation starting at 200 mg QD.
  Other Names: suberoylanilide hydroxamic acid (SAHA)

SUMMARY:
Since the mortality rates for patients with advanced ovarian carinoma are high, the most likely way to improve progression free and overall survival is with maximal "upfront" therapy (Morrow & Curtin, 1998). Currently, no triplet regimen has demonstrated compelling superiority. Therefore, the combination of Paclitaxel, Carboplatin, and Vorinostat is intriguing because of their potential synergy, distinct mechanisms of action, and non-overlapping toxicity.

DETAILED DESCRIPTION:
Ovarian cancer is the fifth most common cancer in women, accounting for nearly 15,280 deaths annually in the United States [1]. Paclitaxel and Carboplatin are currently the accepted standard of care for first line treatment of ovarian cancer [2, 3]. In spite of standard chemotherapy, nearly 70% of patients succumb to this disease. Consequently, studies continue to examine the activity of new agents and dosing regimens to improve disease free intervals and overall survival.

There have been recent data suggesting that weekly chemotherapy regimens may significantly benefit cancer patients' prognosis [4, 5]. Non-small cell lung cancer patient studies employing weekly regimens have shown comparable response and survival rates to Q3 weekly dosing schedules, with a more favorable toxicity profile [6, 7]. Further studies have suggested that weekly Taxane dosing is at least as effective, less toxic, and more convenient than traditional regimens [4, 8, 9].

The favorable activity associated with weekly chemotherapy has primarily been studied in recurrent ovarian cancer patients, investigating the efficacy of single and/or combination drug regimens [10, 11]. However, there have been some studies involving chemo-naïve patients [4, 12, 13]. De Jongh et al. [4} conducted a randomized I/II ovarian cancer trial with cisplatin and escalating doses of weekly or 4-weekly paclitaxel. The chemo-naïve patients exhibited a 94% overall response rate and 48 month median overall survival, while maintaining manageable toxicity. In a more recent advanced ovarian cancer study, Isonishi et al. compared the impact of paclitaxel and carboplatin administered either tri-weekly (c-TC) or dose dense weekly (dd-TC) with regard to patient progression free survival (PFS) [14]. Median PFS for the c-TC patients was 17.1 months and 27.9 months for the dd-TC group. There was also more favorable survival rates in the dose dense patients (83.6%) in comparison to the tri-weekly groups (77.7%)

Shen et al. conducted a Chinese study investigating the efficacy of combination weekly Taxol plus Carboplatin compared to Taxol given every three weeks plus Carboplatin in previously untreated ovarian cancer patients [12]. While the two regimens had equal efficacy, there was less toxicity observed in the weekly regimen. Additional studies have also indicated that lower doses and shorter infusion times inherent in weekly dosing regimens should mitigate bone marrow myelosuppression and other toxicities associated with standard paclitaxel 3-weekly administration [13].

In addition to weekly primary induction chemotherapy regimens, studies involving consolidation or maintenance therapy have been employed in the hopes of improving survival [15, 16]. Micha et al. reported significantly better progression free survival results (94 weeks vs. 45 weeks) for an ovarian cancer group who received 12 cycles of paclitaxel consolidation therapy following induction therapy, compared to a similar group who received 3 cycles of paclitaxel consolidation therapy [16].

The current pilot study was designed to determine toxicity, progression free survival, and response rate of weekly Taxol; every four-week Carboplatin; and Vorinostat (7 days on, 7 days off 7 days on, 7 days off) given for 6 cycles. Some patients will continue on consolidation therapy, which will consist of Taxol in combination with Vorinostat for an additional 12 cycles.

Modifying the dosing schedule of established chemotherapy regimens using weekly chemotherapy administration and consolidation therapy may decrease drug toxicity and maximize efficacy. These benefits are particularly intriguing in patients for whom disease treatment is long-term.

Since no triplet regimen has demonstrated compelling superiority, the combination of Taxol, Carboplatin, and Vorinostat is intriguing because of their potential synergy, distinct mechanisms of action, and non-overlapping toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a histologic or cytologic diagnosis of stage III/IV ovarian cancer, fallopian tube epithelial cancer, or peritoneal cancer who have not received prior chemotherapy or radiotherapy.
* Subjects must have the appropriate surgery for their gynecologic cancer. However, subjects may be treated in a neoadjuvant manner, with surgery being performed after chemotherapy cycles 1, 2, or 3.
* If neoadjuvant therapy is not administered, subjects must receive their first dose no more than six weeks postoperatively.
* Subjects must have adequate bone marrow, renal and hepatic function as defined by WBC > 3,000 cells/cu ml., platelets > 100,000/cu.ml., calculated creatinine clearance > 50 ccs/min., bilirubin < 1.5 mg/dl, and SGOT < three times normal.
* Karnofsky performance status > 50%.
* Subjects who have signed an institutional review board (IRB) approved informed consent form.

Exclusion Criteria:

* Subjects with epithelial ovarian cancer of low malignancy potential.
* Subjects with septicemia, severe infection, or acute hepatitis.
* Subjects with a history of congestive heart failure, angina, or a history of myocardial infarction within the past six months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-10; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Micha, MD, Principal Investigator — Gynecologic Oncology Associates
Locations (1):
- Gynecologic Oncology Associates, Newport Beach, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment was from one location a private practice. The enrollment started on 01/15/2010. The recruitment was to be a two year time period.
Period: Overall Study
Arm/Group | Vorinostat
Started | 18
Completed | 18 (The study was closed on 05/30/12 due to adverse events. We did not complete enrollment)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vorinostat
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 9
Age, Continuous [Median (Full Range); unit: years] | 58 [41 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Clinical response was assessed by clinical, serologic, and radiographic means.
Time Frame: 2 years or 24 months
Population: Response Evaluation Criteria In Solid Tumors (RECIST v1.0)
Measure: Number; unit: participants
Arm/Group | Vorinostat
Number analyzed (Participants) | 18
participants | 12

2. Secondary Outcome: Number of Participants With Progression Free Survival (PFS) up to 24 Months
Description: Progression-free survival was defined as the length of time from the date of initial induction chemotherapy until clinical, radiological, or CA-125 progression
Time Frame: 2 years or 24 months
Measure: Number; unit: participants
Arm/Group | Vorinostat
Number analyzed (Participants) | 18
participants | 18

ADVERSE EVENTS:
Arm/Group | Vorinostat
Serious Adverse Events (participants affected / at risk) | 3/18
Other Adverse Events (participants affected / at risk) | 5/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat (N=18)
gastrointestinal event (Gastrointestinal disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat (N=18)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No